CLINICAL TRIAL: NCT06205732
Title: Retrospective Study and Construction of a Prediction Model for Patients With Intermediate and Advanced Liver Cancer Treated With TACE Combined With Immunotherapy and Targeted Therapy
Brief Title: A Retrospective Study on the Treatment of Intermediate and Advanced Liver Cancer.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: YXLL-KY-2023(145)
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Patient's admission medical records, laboratory tests, etc.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TACE+PD-(L)1+TKI: Application of TACE, TKI, and immunotherapy in patients with intermediate and advanced liver cancer.
  Interventions: Other: Immunotherapy, targeted therapy.
- TACE alone: Application of TACE in patients with intermediate and advanced liver cancer.

INTERVENTIONS:
Other: Immunotherapy, targeted therapy. — Immunotherapy (sintilimab, camrelizumab, tislelizumab, atezolizumab, durvalumab, cardenilumab, and pembrolizumab); targeted therapy (apatinib, lenvatinib, sorafenib, and regorafenib).
  Groups: TACE+PD-(L)1+TKI

SUMMARY:
To evaluate the effectiveness of TACE combined with immunotherapy and targeted therapy versus TACE alone in patients with intermediate and advanced liver cancer.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of TACE combined with immunotherapy and targeted therapy in patients with intermediate and advanced liver cancer. Explore the factors affecting the prognosis of liver cancer treated with TACE combined with immunotherapy and targeted therapy and establish a specific individualized prognostic score and risk stratification model.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old, both men and women
* primary liver cancer confirmed by liver biopsy or history of hepatitis B, AFP, and typical imaging findings
* patients with liver function Child-Pugh A or B (≤8 points)
* BCLC stage B and stage C
* expected survival time ≥8 weeks
* patients with generally good performance status (ECOG PS score 0 or 1)

Exclusion Criteria:

* The patient's key data is missing
* liver metastatic cancer confirmed by histology or cytology
* patients who interrupt treatment due to intolerance of adverse drug reactions
* combined with primary malignant tumors of other organs within 5 years; combined with other serious diseases, such as severe heart disease, renal insufficiency, severe infection, bleeding, etc.
* combined with systemic infection, autoimmune disease, or other types of tumors; previous allogeneic bone marrow transplantation or solid organ transplantation
* study participants known to have mental illness
* situations such as drug use or substance abuse

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with intermediate and advanced liver cancer who received TACE combined with immunotherapy and targeted therapy.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival | 12 months
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Liang, Dr, Study Director — the Qianfoshan Hospital
Locations (1):
- the Qianfoshan Hospital, Jinan, Shandong, China